#### Methods

*Drug.* Capsules containing 500mg Aspirin and identical capsules packed with 500mg microcrystalline cellulose prepared by Pharmacy Specialists (www.makerx.com), a licensed compounding pharmacy.

*Procedure*. Participants will be randomly assigned to either placebo or 500 mg of Aspirin in a double-blind procedure. Participants will fill out background demographic and personality questionnaires for about 20-30 minutes after consuming drug. The tasks will begin after 60 minutes has passed from drug or placebo intake, in order allow sufficient time for Aspirin to be absorbed into the brain (Cryer, 1998; Nagelschmitz, 2014).

Emotional Image Rating Task: Each participant is presented with 120 images, drawn from the previously published stimuli used in Leal et al. (2014), Schaller (2011) and the International Affective Picture System (Lang, 1995), in a pseudo-random order according to the procedures in Durso et al. (2015). Images were pre-categorized on evaluative dimensions corresponding to extremely unpleasant (35 images), moderately unpleasant (15 images), neutral (20 images), moderately pleasant (15 images), and extremely pleasant (35 images). The participants will be asked to evaluate 60 of the images on their valence by being asked the question: "To what extent is this picture positive or negative?" using a 9-point scale with 4 being extremely positive, -4 being extremely negative, and 0 being neither positive nor negative. They will then be shown 60 different images, this time being asked: "To what extent does this picture make you feel an emotional reaction?" in order to rate their level of emotional arousal. A similar 9-point scale was used, with 0 being "I feel little emotion" and 8 being "I feel an extreme amount of emotion." These two blocks are in a consecutive, non-counterbalanced order.

Balloon Analogue Risk Task: Once participants complete the emotional image rating task, they will complete the Balloon Analogue Risk Task (BART) to measure risk taking behavior (Lejuez, et al., 2002). In this task, participants have the opportunity to inflate 15 balloons depicted on the computer screen. A trial begins with a small, uninflated balloon on the computer screen. Participants inflate the balloon, with each pump earning imaginary money, and were told their goal was to earn as much money as possible in the task. Participants could collect their total trial earnings and move them to a permanent bank at any point. However, participants also were told that the balloon can burst as early as the first trial and as late as when the balloon fills the entire computer screen. Bursts were accompanied by a bursting sound and popping animation. If the balloon burst prior to the participants choosing to collect their money, they lost any amount earned thus far on that trial, and had to move on to the next trial having added no money to their permanent bank. Participants were not told about the maximum number of pumps nor the likelihood of bursts, nor that, for each balloon, the first pump had a 1/128 probability of bursting, the second pump 1/127, and so on until on the 128thpump there was a 1/1 probability of bursting.

Memory Recognition Task: Participants are then asked to perform a memory recognition task based on the paradigm in Leal et al. (2014). Participants were shown 180 images and have to classify each as an image that they had seen in the emotional rating task or a new image. Images were divided equally among four different groups: 45 old images that appeared in the emotional rating task, 45 new high similarity lures that looked very closely like images shown in the emotional rating task (ex. an image of a crossing guard, after being shown an image of the same crossing guard from a slightly different angle in the first task), 45 new low similarity lures that looked somewhat like images shown in the emotional rating task (ex. an image of a dirty

Study Design and Analysis Plan: Aspirin Effects on Emotional Reactions, NCT04146532, April 28, 2020 stall, after being shown an image of a dirty toilet in the first task), and 45 new foils that did not bare any resemblance to images from the emotional rating task (ex. an image of an airplane, after not being shown an image of aircraft in the first task). Each group was evenly composed of 9 images from each extremely unpleasant, moderately unpleasant, neutral, moderately pleasant, and extremely pleasant image category. For analysis, d-prime (d') scores were then calculated for each participant in each normative rating category. d' is a measure of a participant's signal detection ability and is unaffected by response bias. It was calculated by subtracting the z-score of each participant's hit rate by the z-score of their false alarm rate for each normative rating category.

Saliva Sample: Participants will then be asked to provide two saliva samples of 1.5 mL in order to measure prostaglandin levels in the saliva. Saliva samples are taken at the beginning of the experiment 5 minutes after the ingestion of drug or placebo, and at the end of the experiment after participants had completed all computerized tasks, approximately 90 minutes after ingestion of drug or placebo.

## **Data Analysis Plan**

For analysis of the evaluations and arousal ratings of the emotional images, identical procedures to those done in Durso, Luttrell, & Way, (2015) will be performed. Specifically, responses will be subjected to a 2 (treatment: Aspirin, placebo) × 5 (normative rating: extremely unpleasant, moderately unpleasant, neutral, moderately pleasant, extremely pleasant) mixed-model ANOVA. Participants who respond faster than 500msec will be dropped from analyses as they are deemed to not be taking the task seriously.

For the Balloon Analogue Risk Task, the primary dependent measure will be adjusted average number of pumps (the number of pumps on trials where the balloon didn't burst) following the initial work in this area (Lejuez, et al., 2002).

For the memory recognition task, the d' score will be subjected to the same analytical approach as that for the evaluations and arousal ratings.

#### References

- Cryer B, Feldman M (1998). Cyclooxygenase-1 and cyclooxygenase-2 selectivity of widely used nonsteroidal anti-inflammatory drugs. *American Journal of Medicine*: 104(5), 413–421. doi: 10.1016/s0002-9343(98)00091-6.
- Durso GRO, Luttrell A, Way BM (2015). Over-the-counter relief from pains and pleasures alike:

  Acetaminophen blunts evaluation sensitivity to both negative and positive stimuli.

  Psychological Science: 26(6), 750–758.
- Hayes, A. F. (2012). PROCESS: A versatile computational tool for observed variable mediation, moderation, and conditional process modeling [White paper]. Retrieved from <a href="http://www.afhayes.com/public/process2012">http://www.afhayes.com/public/process2012</a>.
- Lang P.J. (1995). The Emotion Probe: Studies of Motivation and Attention. *American Psychologist*: 50(5): 372-385.
- Leal S.L., Tighe S.K., Yassa M.A. (2014). Asymmetric effects of emotion on mnemonic interference. *Neurobiol Learn Mem*, 111:41-48.
- Lejuez, C. W., Read J.P., Kahler C.W., Richards J.B., Ramsey S.E., Stuart G.L., Strong D.R., Brown R.A. (2002). Evaluation of a Behavioral Measure of Risk Taking: The Balloon Analogue Risk Task (BART). *Journal of Experimental Psychology: Applied*, 8(2):75–84.
- Nagelschmitz J, Blunck M, Kraetzschmar J, et al (2014). Pharmacokinetics and pharmacodynamics of acetylsalicylic acid after intravenous and oral administration to healthy volunteers. *Clinical Pharmacology*: 6(1), 51–9.

Schaller M., Miller G.E., Gervais W.M., Yager S., Chen E. (2009). Mere Visual Perception of

Other People's Disease Symptoms Facilitates a More Aggressive Immune Response.

Psychological Science: 21(5), 649-652. doi: 10.1177/0956797610368064

# **Appendix**

# Images used in Emotional Image Rating Task

All images from both the emotional image rating task and the memory recognition task were drawn from the previously published stimuli used in Leal et al. (2014), Schaller (2011) and the International Affective Picture System (Lang, 1995). The table below lists the set, image number, and valance category for each image used.

| Image Set | Image Number | Valance Category |
|---|---|---|
| International Affective Picture System | 1052 | Extremely Unpleasant |
| International Affective Picture System | 1111 | Extremely Unpleasant |
| International Affective Picture System | 1201 | Extremely Unpleasant |
| Leal et al. (2014) | 10040a | Extremely Unpleasant |
| Leal et al. (2014) | 10041a | Extremely Unpleasant |
| Leal et al. (2014) | 10044a | Extremely Unpleasant |
| Schaller (2011) | d6 | Extremely Unpleasant |
| Schaller (2011) | d2 | Extremely Unpleasant |
| Schaller (2011) | d4 | Extremely Unpleasant |
| Schaller (2011) | d5 | Extremely Unpleasant |
| Leal et al. (2014) | 10012a | Extremely Unpleasant |
| Leal et al. (2014) | 10023a | Extremely Unpleasant |
| Leal et al. (2014) | 10032a | Extremely Unpleasant |
| Leal et al. (2014) | 10048a | Extremely Unpleasant |
| International Affective Picture System | 6560 | Extremely Unpleasant |
| Leal et al. (2014) | 10035a | Extremely Unpleasant |
| Leal et al. (2014) | 10002a | Extremely Unpleasant |
| Leal et al. (2014) | 10009a | Extremely Unpleasant |
| Leal et al. (2014) | 10025a | Extremely Unpleasant |
| Leal et al. (2014) | 10031a | Extremely Unpleasant |
| Leal et al. (2014) | 10033a | Extremely Unpleasant |
| International Affective Picture System | 3010 | Extremely Unpleasant |
| International Affective Picture System | 3061 | Extremely Unpleasant |
| International Affective Picture System | 3130 | Extremely Unpleasant |
| International Affective Picture System | 3140 | Extremely Unpleasant |
| International Affective Picture System | 3150 | Extremely Unpleasant |
| Leal et al. (2014) | 10038a | Extremely Unpleasant |
| Leal et al. (2014) | 10039a | Extremely Unpleasant |
| Leal et al. (2014) | 10001a | Extremely Unpleasant |
| Leal et al. (2014) | 10010a | Extremely Unpleasant |
| Leal et al. (2014) | 10015a | Extremely Unpleasant |
| Leal et al. (2014) | 10019a | Extremely Unpleasant |
| Leal et al. (2014) | 10020a | Extremely Unpleasant |
| Leal et al. (2014) | 10029a | Extremely Unpleasant |
| Leal et al. (2014) | 10005a | Extremely Unpleasant |
| Schaller (2011) | d10 | Moderately Unpleasant |
| Schaller (2011) | d3 | Moderately Unpleasant |
| International Affective Picture System | 3250 | Moderately Unpleasant |
| International Affective Picture System | 9594 | Moderately Unpleasant |

| Leal et al. (2014) | 10013a | Moderately Unpleasant |
|----------------------------------------|--------|-----------------------|
| Leal et al. (2014) | 10043a | Moderately Unpleasant |
| International Affective Picture System | 2457 | Moderately Unpleasant |
| Leal et al. (2014) | 10022a | Moderately Unpleasant |
| Leal et al. (2014) | 10028a | Moderately Unpleasant |
| Leal et al. (2014) | 10006a | Moderately Unpleasant |
| Leal et al. (2014) | 10016a | Moderately Unpleasant |
| Leal et al. (2014) | 10021a | Moderately Unpleasant |
| Leal et al. (2014) | 10036a | Moderately Unpleasant |
| Leal et al. (2014) | 10045a | Moderately Unpleasant |
| Leal et al. (2014) | 10046a | Moderately Unpleasant |
| Leal et al. (2014) | 20003a | Neutral |
| Leal et al. (2014) | 20010a | Neutral |
| Leal et al. (2014) | 20012a | Neutral |
| Leal et al. (2014) | 20015a | Neutral |
| Leal et al. (2014) | 20016a | Neutral |
| Leal et al. (2014) | 20017a | Neutral |
| Leal et al. (2014) | 20020a | Neutral |
| Leal et al. (2014) | 20022a | Neutral |
| Leal et al. (2014) | 20023a | Neutral |
| Leal et al. (2014) | 20025a | Neutral |
| Leal et al. (2014) | 20026a | Neutral |
| Leal et al. (2014) | 20028a | Neutral |
| Leal et al. (2014) | 20029a | Neutral |
| Leal et al. (2014) | 20031a | Neutral |
| Leal et al. (2014) | 20035a | Neutral |
| Leal et al. (2014) | 20037a | Neutral |
| Leal et al. (2014) | 20038a | Neutral |
| Leal et al. (2014) | 20041a | Neutral |
| Leal et al. (2014) | 20043a | Neutral |
| Leal et al. (2014) | 20048a | Neutral |
| Leal et al. (2014) | 20006a | Moderately Pleasant |
| Leal et al. (2014) | 20007a | Moderately Pleasant |
| Leal et al. (2014) | 20014a | Moderately Pleasant |
| Leal et al. (2014) | 20019a | Moderately Pleasant |
| Leal et al. (2014) | 30009a | Moderately Pleasant |
| Leal et al. (2014) | 30010a | Moderately Pleasant |
| Leal et al. (2014) | 30025a | Moderately Pleasant |
| Leal et al. (2014) | 30030a | Moderately Pleasant |
| Leal et al. (2014) | 30031a | Moderately Pleasant |
| Leal et al. (2014) | 30033a | Moderately Pleasant |
| Leal et al. (2014) | 30034a | Moderately Pleasant |
| Leal et al. (2014) | 30035a | Moderately Pleasant |
| International Affective Picture System | 4800 | Moderately Pleasant |
| Leal et al. (2014) | 30039a | Moderately Pleasant |
| International Affective Picture System | 4647 | Moderately Pleasant |
| International Affective Picture System | 4220 | Extremely Pleasant |
| International Affective Picture System | 4290 | Extremely Pleasant |
| International Affective Picture System | 4660 | Extremely Pleasant |
| International Affective Picture System | 4670 | Extremely Pleasant |
| International Affective Picture System | 4680 | Extremely Pleasant |
| Leal et al. (2014) | 30002a | Extremely Pleasant |
| Leal et al. (2014) | 30003a | Extremely Pleasant |
| 201 00 01. (2011) | 200024 | |

| Leal et al. (2014) | 30005a | Extremely Pleasant |
|--------------------|--------|--------------------|
| Leal et al. (2014) | 30006a | Extremely Pleasant |
| Leal et al. (2014) | 30008a | Extremely Pleasant |
| Leal et al. (2014) | 30011a | Extremely Pleasant |
| Leal et al. (2014) | 30012a | Extremely Pleasant |
| Leal et al. (2014) | 30013a | Extremely Pleasant |
| Leal et al. (2014) | 30015a | Extremely Pleasant |
| Leal et al. (2014) | 30016a | Extremely Pleasant |
| Leal et al. (2014) | 30018a | Extremely Pleasant |
| Leal et al. (2014) | 30019a | Extremely Pleasant |
| Leal et al. (2014) | 30020a | Extremely Pleasant |
| Leal et al. (2014) | 30022a | Extremely Pleasant |
| Leal et al. (2014) | 30023a | Extremely Pleasant |
| Leal et al. (2014) | 30026a | Extremely Pleasant |
| Leal et al. (2014) | 30027a | Extremely Pleasant |
| Leal et al. (2014) | 30028a | Extremely Pleasant |
| Leal et al. (2014) | 30029a | Extremely Pleasant |
| Leal et al. (2014) | 30036a | Extremely Pleasant |
| Leal et al. (2014) | 30040a | Extremely Pleasant |
| Leal et al. (2014) | 30041a | Extremely Pleasant |
| Leal et al. (2014) | 30042a | Extremely Pleasant |
| Leal et al. (2014) | 30045a | Extremely Pleasant |
| Leal et al. (2014) | 30046a | Extremely Pleasant |
| Leal et al. (2014) | 30047a | Extremely Pleasant |
| Leal et al. (2014) | 30049a | Extremely Pleasant |
| Leal et al. (2014) | 30051a | Extremely Pleasant |
| Leal et al. (2014) | 30050a | Extremely Pleasant |
| - | | - |

# Images used in Memory Recognition Task

| Image Set | Image Number | Valance Category | Target/Foil/Lure |
|---|---|---|---|
| Leal et. al (2014) | 10012a | Extremely Unpleasant | Target |
| Leal et. al (2014) | 10039a | Extremely Unpleasant | Target |
| Leal et. al (2014) | 10041a | Extremely Unpleasant | Target |
| Leal et. al (2014) | 10009a | Extremely Unpleasant | Target |
| Leal et. al (2014) | 10015a | Extremely Unpleasant | Target |
| Schaller (2012) | d6 | Extremely Unpleasant | Target |
| Schaller (2012) | d5 | Extremely Unpleasant | Target |
| International Affective Picture System | 6560 | Extremely Unpleasant | Target |
| Leal et. al (2014) | 10005a | Extremely Unpleasant | Target |
| Leal et. al (2014) | 10043a | Moderately Unpleasant | Target |
| Leal et. al (2014) | 10046a | Moderately Unpleasant | Target |
| Leal et. al (2014) | 10022a | Moderately Unpleasant | Target |
| Leal et. al (2014) | 10013a | Moderately Unpleasant | Target |
| Leal et. al (2014) | 10016a | Moderately Unpleasant | Target |
| Leal et. al (2014) | 10036a | Moderately Unpleasant | Target |
| Schaller (2012) | d3 | Moderately Unpleasant | Target |
| Schaller (2012) | d10 | Moderately Unpleasant | Target |
| International Affective Picture System | 2457 | Moderately Unpleasant | Target |
| Leal et. al (2014) | 20029a | Neutral | Target |
| Leal et. al (2014) | 20026a | Neutral | Target |
| Leal et. al (2014) | 20025a | Neutral | Target |
| Leal et. al (2014) | 20028a | Neutral | Target |
| Leal et. al (2014) | 20022a | Neutral | Target |
| Leal et. al (2014) | 20003a | Neutral | Target |
| Leal et. al (2014) | 20010a | Neutral | Target |
| Leal et. al (2014) | 20012a | Neutral | Target |
| Leal et. al (2014) | 20017a | Neutral | Target |
| International Affective Picture System | 4647 | Moderately Pleasant | Target |
| Leal et. al (2014) | 30034a | Moderately Pleasant | Target |
| International Affective Picture System | 4800 | Moderately Pleasant | Target |
| Leal et. al (2014) | 30035a | Moderately Pleasant | Target |
| Leal et. al (2014) | et. al (2014) 30010a Moderately Pleasant | | Target |
| Leal et. al (2014) | 20007a | Moderately Pleasant | Target |
| Leal et. al (2014) | 20006a | Moderately Pleasant | Target |
| Leal et. al (2014) | 30009a | Moderately Pleasant | Target |
| Leal et. al (2014) | 30030a | Moderately Pleasant | Target |
| International Affective Picture System | 4220 | Extremely Pleasant | Target |
| Leal et. al (2014) | 30003a | Extremely Pleasant | Target |
| International Affective Picture System | 4660 | Extremely Pleasant | Target |
| Leal et. al (2014) | 30051a | Extremely Pleasant | Target |
| International Affective Picture System | 4290 | Extremely Pleasant | Target |
| Leal et. al (2014) | 30012a | Extremely Pleasant | Target |
| International Affective Picture System | 4670 | Extremely Pleasant | Target |
| Leal et. al (2014) | 30018a | Extremely Pleasant | Target |
| Leal et. al (2014) | 30019a | Extremely Pleasant | Target |
| Leal et. al (2014) | 10023c | Extremely Unpleasant | High Similarity Lure |
| Leal et. al (2014) | 10005c | Extremely Unpleasant | High Similarity Lure |
| Leal et. al (2014) | 10035c | Extremely Unpleasant | High Similarity Lure |
| Leal et. al (2014) | 10002c | Extremely Unpleasant | High Similarity Lure |

| Loglot al (2014) | 10021. | Entrare de Harles sont | High Cincilonity Lynn |
|---|---|---|---|
| Leal et. al (2014) | 10031c | Extremely Unpleasant | High Similarity Lure |
| Leal et. al (2014) | 10001c | Extremely Unpleasant | High Similarity Lure |
| Leal et. al (2014) | 10038c | Extremely Unpleasant | High Similarity Lure |
| Leal et. al (2014) | 10029c | Extremely Unpleasant | High Similarity Lure |
| Leal et. al (2014) | 10025c | Extremely Unpleasant | High Similarity Lure |
| Leal et. al (2014) | 10043c | Moderately Unpleasant | High Similarity Lure |
| Leal et. al (2014) | 10013c | Moderately Unpleasant | High Similarity Lure |
| Leal et. al (2014) | 10046c | Moderately Unpleasant | High Similarity Lure |
| Leal et. al (2014) | 10045c | Moderately Unpleasant | High Similarity Lure |
| Leal et. al (2014) | 10021c | Moderately Unpleasant | High Similarity Lure |
| Leal et. al (2014) | 10022c | Moderately Unpleasant | High Similarity Lure |
| Leal et. al (2014) | 10046c | Moderately Unpleasant | High Similarity Lure |
| Leal et. al (2014) | 10036c | Moderately Unpleasant | High Similarity Lure |
| Leal et. al (2014) | 10006c | Moderately Unpleasant | High Similarity Lure |
| Leal et. al (2014) | 20037c | Neutral | High Similarity Lure |
| Leal et. al (2014) | 20029c | Neutral | High Similarity Lure |
| Leal et. al (2014) | 20025c | Neutral | High Similarity Lure |
| Leal et. al (2014) | 20043c | Neutral | High Similarity Lure |
| Leal et. al (2014) | 20031c | Neutral | High Similarity Lure |
| Leal et. al (2014) | 20035c | Neutral | High Similarity Lure |
| Leal et. al (2014) | 20003c | Neutral | High Similarity Lure |
| Leal et. al (2014) | 20010c | Neutral | High Similarity Lure |
| Leal et. al (2014) | 20015c | Neutral | High Similarity Lure |
| Leal et. al (2014) | 20019c | Moderately Pleasant | High Similarity Lure |
| Leal et. al (2014) | 30034c | Moderately Pleasant | High Similarity Lure |
| Leal et. al (2014) | 20014c | Moderately Pleasant | High Similarity Lure |
| Leal et. al (2014) | 30033c | Moderately Pleasant | High Similarity Lure |
| Leal et. al (2014) | 30039c | Moderately Pleasant | High Similarity Lure |
| Leal et. al (2014) | 30035c | Moderately Pleasant | High Similarity Lure |
| Leal et. al (2014) | 20006c | Moderately Pleasant | High Similarity Lure |
| Leal et. al (2014) | 30009c | Moderately Pleasant | High Similarity Lure |
| Leal et. al (2014) | 30010c | Moderately Pleasant | High Similarity Lure |
| Leal et. al (2014) | 30019c | Extremely Pleasant | High Similarity Lure |
| Leal et. al (2014) | 30013c | Extremely Pleasant | High Similarity Lure |
| Leal et. al (2014) | 30016c | Extremely Pleasant | High Similarity Lure |
| Leal et. al (2014) | 30023c | Extremely Pleasant | High Similarity Lure |
| Leal et. al (2014) | 30046c | Extremely Pleasant | High Similarity Lure |
| Leal et. al (2014) | 30008c | Extremely Pleasant | High Similarity Lure |
| Leal et. al (2014) | 30002c | Extremely Pleasant | High Similarity Lure |
| Leal et. al (2014) | 30005c | Extremely Pleasant | High Similarity Lure |
| Leal et. al (2014) | 30020c | Extremely Pleasant | High Similarity Lure |
| Leal et. al (2014) | 10032b | Extremely Unpleasant | Low Similarity Lure |
| Leal et. al (2014) | 10039b | Extremely Unpleasant | Low Similarity Lure |
| Leal et. al (2014) | 10048b | Extremely Unpleasant | Low Similarity Lure |
| Leal et. al (2014) | 10031b | Extremely Unpleasant | Low Similarity Lure |
| Leal et. al (2014) | 10040b | Extremely Unpleasant | Low Similarity Lure |
| Leal et. al (2014) | 10020b | Extremely Unpleasant | Low Similarity Lure |
| Leal et. al (2014) | 10012b | Extremely Unpleasant | Low Similarity Lure |
| Leal et. al (2014) | 10023b | Extremely Unpleasant | Low Similarity Lure |
| Leal et. al (2014) | 10035b | Extremely Unpleasant | Low Similarity Lure |
| Leal et. al (2014) | 10013b | Moderately Unpleasant | Low Similarity Lure |
| Leal et. al (2014) | 10036b | Moderately Unpleasant | Low Similarity Lure |
| Leal et. al (2014) | 10006b | Moderately Unpleasant | Low Similarity Lure |
| Dour Ot. ar (2017) | 100000 | into del atery empreusum | 2011 Similarity Duit |

| I and at al (2014) | 10017 | Moderately Huntagent | I am Cincilanita I ama |
|--------------------|--------|-----------------------|------------------------|
| Leal et. al (2014) | 10016b | Moderately Unpleasant | Low Similarity Lure |
| Leal et. al (2014) | 10021b | Moderately Unpleasant | Low Similarity Lure |
| Leal et. al (2014) | 10028b | Moderately Unpleasant | Low Similarity Lure |
| Leal et. al (2014) | 10043b | Moderately Unpleasant | Low Similarity Lure |
| Leal et. al (2014) | 10022b | Moderately Unpleasant | Low Similarity Lure |
| Leal et. al (2014) | 10046b | Moderately Unpleasant | Low Similarity Lure |
| Leal et. al (2014) | 20048b | Neutral | Low Similarity Lure |
| Leal et. al (2014) | 20026b | Neutral | Low Similarity Lure |
| Leal et. al (2014) | 20025b | Neutral | Low Similarity Lure |
| Leal et. al (2014) | 20022b | Neutral | Low Similarity Lure |
| Leal et. al (2014) | 20017b | Neutral | Low Similarity Lure |
| Leal et. al (2014) | 20016b | Neutral | Low Similarity Lure |
| Leal et. al (2014) | 20003b | Neutral | Low Similarity Lure |
| Leal et. al (2014) | 20010b | Neutral | Low Similarity Lure |
| Leal et. al (2014) | 20012b | Neutral | Low Similarity Lure |
| Leal et. al (2014) | 30010b | Moderately Pleasant | Low Similarity Lure |
| Leal et. al (2014) | 20006b | Moderately Pleasant | Low Similarity Lure |
| Leal et. al (2014) | 30030b | Moderately Pleasant | Low Similarity Lure |
| Leal et. al (2014) | 20007b | Moderately Pleasant | Low Similarity Lure |
| Leal et. al (2014) | 20014b | Moderately Pleasant | Low Similarity Lure |
| Leal et. al (2014) | 30031b | Moderately Pleasant | Low Similarity Lure |
| Leal et. al (2014) | 30009b | Moderately Pleasant | Low Similarity Lure |
| Leal et. al (2014) | 30033b | Moderately Pleasant | Low Similarity Lure |
| Leal et. al (2014) | 30035b | Moderately Pleasant | Low Similarity Lure |
| Leal et. al (2014) | 30003b | Extremely Pleasant | Low Similarity Lure |
| Leal et. al (2014) | 30011b | Extremely Pleasant | Low Similarity Lure |
| Leal et. al (2014) | 30040b | Extremely Pleasant | Low Similarity Lure |
| Leal et. al (2014) | 30049b | Extremely Pleasant | Low Similarity Lure |
| Leal et. al (2014) | 30018b | Extremely Pleasant | Low Similarity Lure |
| Leal et. al (2014) | 30029b | Extremely Pleasant | Low Similarity Lure |
| Leal et. al (2014) | 30002b | Extremely Pleasant | Low Similarity Lure |
| Leal et. al (2014) | 30036b | Extremely Pleasant | Low Similarity Lure |
| Leal et. al (2014) | 30026b | Extremely Pleasant | Low Similarity Lure |
| Leal et. al (2014) | 40041a | Extremely Unpleasant | Foil |
| Leal et. al (2014) | 40038a | Extremely Unpleasant | Foil |
| Leal et. al (2014) | 40006a | Extremely Unpleasant | Foil |
| Leal et. al (2014) | 40009a | Extremely Unpleasant | Foil |
| Leal et. al (2014) | 40022a | Extremely Unpleasant | Foil |
| Leal et. al (2014) | 40035a | Extremely Unpleasant | Foil |
| Leal et. al (2014) | 40002a | Extremely Unpleasant | Foil |
| Leal et. al (2014) | 40010a | Extremely Unpleasant | Foil |
| Leal et. al (2014) | 40011a | Extremely Unpleasant | Foil |
| Leal et. al (2014) | 40007a | Moderately Unpleasant | Foil |
| Leal et. al (2014) | 40013a | Moderately Unpleasant | Foil |
| Leal et. al (2014) | 40028a | Moderately Unpleasant | Foil |
| Leal et. al (2014) | 40031a | Moderately Unpleasant | Foil |
| Leal et. al (2014) | 40044a | Moderately Unpleasant | Foil |
| Leal et. al (2014) | 40029a | Moderately Unpleasant | Foil |
| Leal et. al (2014) | 40008a | Moderately Unpleasant | Foil |
| Leal et. al (2014) | 40012a | Moderately Unpleasant | Foil |
| Leal et. al (2014) | 40015a | Moderately Unpleasant | Foil |
| Leal et. al (2014) | 50005a | Neutral | Foil |
| Leal et. al (2014) | 50007a | Neutral | Foil |
| Loai ot. ai (2014) | 30007a | redual | 1 011 |

Study Design and Analysis Plan: Aspirin Effects on Emotional Reactions, NCT04146532, April 28, 2020

| | ı | |
|---|---|---|
| 50010a | Neutral | Foil |
| 50014a | Neutral | Foil |
| 50016a | Neutral | Foil |
| 50042a | Neutral | Foil |
| 50013a | Neutral | Foil |
| 50017a | Neutral | Foil |
| 50018a | Neutral | Foil |
| 60001a | Moderately Pleasant | Foil |
| 60003a | Moderately Pleasant | Foil |
| 60011a | Moderately Pleasant | Foil |
| 60019a | Moderately Pleasant | Foil |
| 60002a | Moderately Pleasant | Foil |
| 60004a | Moderately Pleasant | Foil |
| 60017a | Moderately Pleasant | Foil |
| 60032a | Moderately Pleasant | Foil |
| 60041a | Moderately Pleasant | Foil |
| 60048a | Extremely Pleasant | Foil |
| 60043a | Extremely Pleasant | Foil |
| 60038a | Extremely Pleasant | Foil |
| 60033a | Extremely Pleasant | Foil |
| 60027a | Extremely Pleasant | Foil |
| 60010a | Extremely Pleasant | Foil |
| 60039a | Extremely Pleasant | Foil |
| 60024a | Extremely Pleasant | Foil |
| 60020a | Extremely Pleasant | Foil |
| | 50016a<br>50042a<br>50013a<br>50017a<br>50018a<br>60001a<br>60003a<br>60011a<br>60019a<br>60002a<br>60004a<br>60017a<br>60032a<br>60041a<br>60048a<br>60048a<br>60038a<br>60038a<br>60027a<br>60010a<br>60039a<br>60024a | 50014a Neutral 50016a Neutral 50042a Neutral 50013a Neutral 50017a Neutral 50018a Neutral 60001a Moderately Pleasant 60003a Moderately Pleasant 60011a Moderately Pleasant 60019a Moderately Pleasant 60002a Moderately Pleasant 60004a Moderately Pleasant 60017a Moderately Pleasant 60032a Moderately Pleasant 60041a Moderately Pleasant 60048a Extremely Pleasant 60038a Extremely Pleasant 60033a Extremely Pleasant 60027a Extremely Pleasant 60010a Extremely Pleasant 60039a Extremely Pleasant 60024a Extremely Pleasant |

# Questionnaires

# Background Measures Recent Health Behaviors Questionnaire

| 1. | What is your height?feetinches |
|---|---|
| 2. | What is your weight? (in pounds) |
| 3. | What time did you go to bed last night? |
| 4. | How long (in minutes) did it take you to fall asleep last night? |
| 5. | What time did you get up this morning? |
| 6. | On a scale of 1 to 10, how well did you sleep? (1=poorly, 10=well) |
| 7. | How many hours of actual sleep did you get? (This may be different than the number of hours you spent in bed? |
| 8. | Approximately how long ago did you last eat? Was it a (indicate one): Snack Light Meal Full Meal |
| 9. | Have you done any aerobic exercise today? If yes, how many minutes? If yes, how long ago (in hours)? |
| 10. | On an average week, how many days do you do aerobic exercise? |

| 11. | When you do exercise, how long do you usually work out? (in minutes) | | | | | |
|---|---|---|---|---|---|---|
| 1. | In general, would you sa | y that your health | is (indicate | e one): | | |
| | Excellent Very Go | od Good | Fa | ir | Poor | |
| 1 | Please answer the following 3 questions by circling a number on the right: | Strongly<br>Disagree | | | | Strongly<br>Agree |
| 2. | Over the last couple of days, I have not been feeling well. | 1 | 2 | 3 | 4 | 5 |
| 3. | Lately, I have been feeling a little under the weather | 1 | 2 | 3 | 4 | 5 |
| 4. | I have felt sick within the last week. | 1 | 2 | 3 | 4 | 5 |
| 5. | When was the last time you had a cold, flu, dental infection, or other infection? Today A couple of days ago A week ago A couple of weeks ago A month ago A few months ago A year or more ago | | | | | |
| 6. | Did you seek medical ca<br>No | · | | | | |
| | If yes, how many times i illness? | n the last 3 month | | | aith center | ior an |
| 7. | Did you take any over-th<br>No<br>any infection in the last | · | cription me | edications f | or a cold, fl | u, or Yes |

| | If yes, what medications |
|---|---|
| | Please answer the following questions by circling a response on the right: |
| | 1. In the box below, please list all medications AND vitamins or supplements you are currently taking, including pills, patches, lotions or injections. Medications can be prescription medications or over-the-counter medications. Be sure to include the NAME, DOSE, AMOUNT and FREQUENCY you take the medications or supplements, putting a comma between each one. If the medication or supplement does not have a particular dose, please put "NA" after name and before frequency. See examples below. |
| | Example 1: Oxytrol 3.9 mg 1 patch every 4 days, Femgest progesterone cream no dosage apply to hands once per day, Synthroid 75 mcg 1 pill once per day. |
| | Example 2: Timoptic 0.25% 2 drops per eye twice per day, Saw Palmetto 160 mg 1 pill twice per day, Zocor 20 mg each night. |
| | Example 3: Calcium 333mg/pill 3 pills per day, Vitamin C 500mg 1 pill per day, Vitamin D 1000mg 1 pill per day. |
| 2. | Are you currently taking birth control medication? Yes No |
| 3. | How often do you typically use marijuana? (indicate one) |
| | Almost every day At least once a month |
| | Several times a week Several times a year |
| | At least once a week At least once a year |

| | Several t | times a month | | Never | | |
|---|---|---|---|---|---|---|
| 4. | | = | e marijuana? (If i<br>per of days, mont | n the last day, ple<br>hs, or years.) | ase indicate the I | number of |
| | Hours: | Days: | Month | ıs: Ye | ears: | - |
| | I have | never used mari | juana. | | | |
| 5. | How many c | igarettes per day | do you smoke (i | ndicate one respo | nse)? | |
| | 0 | 1 to 10 | 10 to 20 2 | 0 to 30 30 o | r more | |
| 6. | If you smoke<br>minutes and | <del>-</del> | been since your | last cigarette? (Pl | ease indicate the | number of |
| | | Minutes: | Hours: | <u> </u> | | |
| 7. | . When was the last time you consumed an alcoholic beverage? (If in the last day, please indicate the number of hours. If not record the number of days, months, or years.) | | | | | |
| | Hours: | Days: | Month | s: Ye | ears: | - |
| | I do no | ot drink alcohol. | | | | |
| | Please answer the | following 3 que | stions by circling | a response on the | e right: | |
| | How | | , , | 2 - 4 times a | 2-3 | 4 or more |
| 8. | often do<br>you have<br>a drink<br>containing<br>alcohol? | Never | Monthly | month | times a<br>week | times a week |
| 9. | How many drinks containing alcohol do you have on a typical | 1 or 2 | 3 or 4 | 5 or 6 | 7 to 9 | 10 or<br>more |

| | day when<br>you are<br>drinking? | | | | | | |
|---|---|---|---|---|---|---|---|
| 10. | How often do you have six or more drinks on one occasion? | Never | Less<br>than<br>Monthly | Monthly | , | Weekly | Daily or<br>almost<br>Daily |
| | | | l | | | | |
| 11. | Do you have a | rthritis, rheumat | oid arthritis, or joi | int problems? | Υe | es 1 | No |
| 12. | <del>-</del> | rthritis or any im<br>ency such as HIV? | mune disorders th | nat might lead to | o<br>Yes | No | |
| 13. | | ny chronic illness<br>em (e.g Cushing' | ses that affect the ss Disease)? | | Yes | No | |
| 14. | Are you diabet | ic (Type I or II)? | | | Yes | No | |

# Think of this ladder as representing where people stand in the United States.

At the **top** of the ladder are the people who are best off—those who have the most money, the most education, and the most respected jobs. At the **bottom** are the people who are the worst off— who have the least money, least education, and the least respected jobs or no job. The higher up you are on this ladder, the closer you are to the people at the very top; the lower you are, the closer you are to the people at the very bottom.

# Where would you place yourself on this ladder?

Please place a large "X" on the rung where you think you stand at this time in your life, relative to other people in the United States.



# Political Ideology (Wilson, 1968)

G.D. Wilson, J.R. Patterson, A new measure of conservatism, Br. J. Soc. Clin.Psychol. 7 (1968) 264–269. Mofied by Mills, M., Gonzalez, F. J., Giuseffi, K., Sievert, B., Smith, K. B., Hibbing, J. R., & Dodd, M. D. (2016). Political conservatism predicts asymmetries in emotional scene memory. *Behavioural brain research*, 306, 84–90.

Indicate your agreement with the following issues:

| , , | strongly<br>disagree with<br>(1) | disagree with (2) | uncertain<br>about (3) | agree with (4) | strongly agree<br>with (5) |
|---|---|---|---|---|---|
| school prayer (1) | $\circ$ | $\circ$ | $\circ$ | $\bigcirc$ | $\bigcirc$ |
| pacifism (2) | | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ |
| stopping immigration (3) | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| death penalty<br>(4) | $\circ$ | $\circ$ | $\circ$ | $\circ$ | $\circ$ |
| government-<br>arranged<br>healthcare (5) | $\circ$ | $\circ$ | $\circ$ | $\circ$ | 0 |
| premarital sex<br>(6) | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ |
| gay marriage<br>(7) | $\bigcirc$ | $\circ$ | $\bigcirc$ | $\circ$ | $\bigcirc$ |
| abortion rights (8) | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ |
| evolution (9) | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ |
| biblical truth<br>(10) | $\circ$ | $\bigcirc$ | $\circ$ | $\circ$ | $\bigcirc$ |
| increased<br>welfare<br>spending (11) | 0 | 0 | 0 | $\circ$ | 0 |
| protecting gun rights (12) | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ | $\bigcirc$ |
| increasing<br>military<br>spending (13) | 0 | 0 | $\circ$ | $\circ$ | $\circ$ |
| government<br>regulation of<br>business (14) | $\bigcirc$ | 0 | $\circ$ | $\circ$ | $\circ$ |
| small<br>government<br>(15) | 0 | $\circ$ | $\circ$ | $\circ$ | $\circ$ |

| Study Design an | d Analysis Pla | n: Aspirin Effec | ts on Emotiona | Reactions, NCT | 04146532, April 2 | 8, 2020 |
|---|---|---|---|---|---|---|
| foreign aide<br>(16) | $\circ$ | $\circ$ | | | 0 | $\circ$ |
| lowering taxe (17) | S | $\circ$ | | | 0 | $\bigcirc$ |
| stem cell<br>research (18) | $\bigcirc$ | $\circ$ | | | 0 | $\bigcirc$ |
| abstinence-<br>only sex<br>education (19 | () | $\circ$ | | | 0 | $\bigcirc$ |
| allowing<br>torture of<br>terrorism<br>suspects (20) | 0 | 0 | | | 0 | 0 |
| When it comes to politics in general, do you usually think of yourself as liberal, moderate, or conservative? | | | | | | |
| O very libera | l (1) | | | | | |
| O liberal (2) | | | | | | |
| osomewhat | liberal (3) | | | | | |
| O moderate | (4) | | | | | |
| osomewhat | conservative | (5) | | | | |
| O conservati | ve (6) | | | | | |
| O very conse | rvative (7) | | | | | |
| In general, I co | nsider myself | a: | | | | |
| O Democrat | (1) | | | | | |
| O Republicar | n (2) | | | | | |
| OLibertarian | (3) | | | | | |
| Other (4) | | | | | | |
| When it comes or something e | | general, do yo | ou usually thin | k of yourself as I | iberal, moderat | e, conservative |
| Very<br>Liberal<br>1 | Liberal<br>2 | Somewhat<br>Liberal<br>3 | Moderate<br>4 | Somewhat<br>Conservative<br>5 | Conservative<br>6 | Very<br>Conservative<br>7 |

On social issues, you consider yourself to be:

| Very | | Somewhat | | Somewhat | Very | |
|---|---|---|---|---|---|---|
| Liberal | Liberal | Liberal | Moderate | Conservative | Conservative | Conservative |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 |

On foreign policy issues, you consider yourself to be:

| Very | | Somewhat | | Somewhat | Very | |
|---|---|---|---|---|---|---|
| Liberal | Liberal | Liberal | Moderate | Conservative | Conservative | Conservative |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 |

On economic issues, you consider yourself to be:

| Very | | Somewhat | | Somewhat | Very | |
|---|---|---|---|---|---|---|
| Liberal | Liberal | Liberal | Moderate | Conservative | Conservative | Conservative |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 |

#### **Emotionality Measures**

Domain Specific Risk Taking (Blais & Weber, 2006)

Blais, A. & Weber, E. U. (2006). A domain-specific risk-taking (DOSPERT) scale for adult populations. *Judgment and Decision Making*, 1(1): 33-47.

#### **Risk Perception**

People often see some risk in situations that contain uncertainty about what the outcome or consequences will be and for which there is the possibility of negative consequences. However, riskiness is a very personal and intuitive notion, and we are interested in your gut level assessment of how risky each situation or behavior is. For each of the following statements, please indicate how risky you perceive each situation. Provide a rating from Not at all Risky to Extremely Risky, using the following scale:

1 Not at all Risky 2 Slightly Risky 3 Somewhat Risky 4 Moderately Risky 5 Risky 6 Very Risky 7Extremely Risky

#### **Expected Benefits**

For each of the following statements, please indicate the benefits you would obtain from each situation. Provide a rating from 1 to 7, using the following scale:

1 No Benefits at all 2 3 4 Moderate Benefits 5 6 7 Great Benefits

#### **Items**

- 1. Admitting that your tastes are different from those of a friend. (S)
- 2.Going camping in the wilderness. (R)
- 3.Betting a day's income at the horse races. (F/G)
- 4.Investing 10% of your annual income in a moderate growth diversified fund. (F/I)
- 5. Drinking heavily at a social function. (H/S)
- 6. Taking some questionable deductions on your income tax return. (E)
- 7. Disagreeing with an authority figure on a major issue. (S)
- 8.Betting a day's income at a high-stake poker game. (F/G)
- 9. Having an affair with a married man/woman. (E)
- 10. Passing off somebody else's work as your own. (E)
- 11. Going down a ski run that is beyond your ability. (R)
- 12. Investing 5% of your annual income in a very speculative stock. (F/I)

- 13. Going whitewater rafting at high water in the spring. (R)
- 14.Betting a day's income on the outcome of a sporting event (F/G)
- 15.Engaging in unprotected sex. (H/S)
- 16. Revealing a friend's secret to someone else. (E)
- 17. Driving a car without wearing a seat belt. (H/S)
- 18.Investing 10% of your annual income in a new business venture. (F/I)
- 19. Taking a skydiving class. (R)
- 20. Riding a motorcycle without a helmet. (H/S)
- 21. Choosing a career that you truly enjoy over a more secure one. (S)
- 22. Speaking your mind about an unpopular issue in a meeting at work. (S)
- 23. Sunbathing without sunscreen. (H/S)
- 24.Bungee jumping off a tall bridge. (R)
- 25. Piloting a small plane. (R)
- 26. Walking home alone at night in an unsafe area of town. (H/S)
- 27. Moving to a city far away from your extended family. (S)
- 28. Starting a new career in your mid-thirties. (S)
- 29.Leaving your young children alone at home while running an errand. (E)
- 30. Not returning a wallet you found that contains \$200. (E)

*Note*. E = Ethical, F = Financial, H/S = Health/Safety, R = Recreational, and S = Social.

### Toronto Alexithymia Scale

Bagby, R. M., Parker, J. D. A. & Taylor, G. J. (1994). The twenty-item Toronto Alexithymia Scale-I. Item selection and cross-validation of the factor structure. Journal of Psychosomatic Research, 38, 23-32.

# TAS - 20

Using the scale provided as a guide, indicate how much you agree or disagree with each of the following statements by circling the appropriate number. Circle only one number for each statement.

1 = STRONGLY DISAGREE

- 2 = MODERATELY DISAGREE
- 3 = NEITHER DISAGREE NOR AGREE
- 4 = MODERATELY AGREE
- 5 = STRONGLY AGREE

| 1. | I am often confused about what emotion I am feeling. | 1. | 1 | 2 | 3 | 4 | 5 |
|---|---|---|---|---|---|---|---|
| 2. | It is difficult for me to find the right words for my | 2. | 1 | 2 | 3 | 4 | 5 |
| | feelings. | | | | | | |
| 3. | I have physical sensations that even doctors don't | 3. | 1 | 2 | 3 | 4 | 5 |
| | understand. | | | | | | |
| 4. | I am able to describe my feelings easily. | 4. | 1 | 2 | 3 | 4 | 5 |
| 5. | I prefer to analyze problems rather than just describe | 5. | 1 | 2 | 3 | 4 | 5 |
| | them. | | | | | | |
| 6. | When I am upset, I don't know if I am sad, frightened, or | 6. | 1 | 2 | 3 | 4 | 5 |
| | angry. | | | | | | |
| 7. | I am often puzzled by sensations in my body. | 7. | 1 | 2 | 3 | 4 | 5 |
| 8. | I prefer to just let things happen rather than to understand | 8. | 1 | 2 | 3 | 4 | 5 |
| | why they turned out that way. | 9. | 1 | 2 | 3 | 4 | 5 |
| 9. | I have feelings that I can't quite identify. | 10. | 1 | 2 | 3 | 4 | 5 |
| 10. | Being in touch with emotions is essential. | | | | | | |
| 11. | I find it hard to describe how I feel about people. | 11. | 1 | 2 | 3 | 4 | 5 |
| 12. | People tell me to describe my feelings more. | 12. | 1 | 2 | 3 | 4 | 5 |
| 13. | I don't know what's going on inside me. | 13. | 1 | 2 | 3 | 4 | 5 |
| 14. | I often don't know why I am angry. | 14. | 1 | 2 | 3 | 4 | 5 |
| 15. | I prefer talking to people about their daily activities rather | 15. | 1 | 2 | 3 | 4 | 5 |
| | than their feelings | | | | | | |
| 16. | I prefer to watch "light" entertainment shows rather than | 16. | 1 | 2 | 3 | 4 | 5 |
| | psychological dramas. | | | | | | |
| 17. | It is difficult for me to reveal my innermost feelings, even | 17. | 1 | 2 | 3 | 4 | 5 |
| | to close friends. | | | | | | |
| 18. | I can feel close to someone, even in moments of silence. | 18. | 1 | 2 | 3 | 4 | 5 |
| 19. | I find examination of my feelings useful in solving | 19. | 1 | 2 | 3 | 4 | 5 |
| | personal problems. | | | | | | |
| 20. | Looking for hidden meanings in movies or plays distracts | 20. | 1 | 2 | 3 | 4 | 5 |
| | from their enjoyment. | | | | | | |

#### Highly Sensitive Persons Scale (Pluess, 2018)

Pluess, M., Assary, E., Lionetti, F., Lester, K. J., Krapohl, E., Aron, E. N., & Aron, A. (2018). Environmental sensitivity in children: Development of the Highly Sensitive Child Scale and identification of sensitivity groups. *Developmental psychology*, 54(1), 51.

- 1. I find it unpleasant to have a lot going on at once
- 2. Some music can make me really happy
- 3. I love nice tastes
- 4. Loud noises make me feel uncomfortable
- 5. I am annoyed when people try to get me to do too many things at once
- 6. I notice it when small things have changed in my environment
- 7. I get nervous when I have to do a lot in little time
- 8. I love nice smells
- 9. I don't like watching TV programs that have a lot of violence in them
- 10. I don't like loud noises
- 11. I don't like it when things change in my life
- 12 When someone observes me, I get nervous. This makes me perform worse than normal.

The Positive and Negative Affectivity Scale Questionnaire (PANAS; Watson, Clark, & Tellegan, 1988)

Watson D., Clark, L. A., & Tellegan, A. (1988). Development and validation of brief measures of positive and negative affect: The PANAS scales. *Journal of Personality and Social Psychology*, 54(6): 1063-1070.

This scale consists of a number of words that describe different feelings and emotions. Read each item and then list the number from the scale below next to each word. Indicate to what extent you feel this way right now, that is, at the present moment OR indicate the extent you have felt this way over the past week (circle the instructions you followed when taking this measure)

| Very Slightly or Not at All | A Little | | Moderately | Quite a Bit | Extremely |
|---|---|---|---|---|---|
| 1 | 2 | 3 | 4 | | 5 |
| 1. Interested | | = | 11. Irrit | able | |
| 2. Distressed | | - | 12. Aler | t | |
| 3. Excited | | = | 13. Ash | amed | |
| 4. Upset | | _ | 14. Insp | oired | |
| 5. Strong | | _ | 15. Ner | vous | |
| 6. Guilty | | _ | 16. Det | ermined | |
| 7. Scared | | _ | 17. Atte | entive | |
| 8. Hostile | | _ | 18. Jitte | ery | |
| 9. Enthusiastic | | _ | 19. Acti | ve | |
| 10. Proud | | _ | 20. Afra | nid | |

# Tybur 3 Domain Disgust Questionnaire (Tybur, 2009)

Tybur, J. M., Lieberman, D., & Griskevicius, V. (2009). Microbes, mating, and morality: Individual differences in three functional domains of disgust. *Journal of Personality and Social Psychology*, *97*: 103–122.

The following items describe a variety of concepts. Please rate how disgusting you find the concepts described in the items, where 0 means that you do not find the concept disgusting at all and 6 means that you find the concept extremely disgusting.

| | Not at all<br>disgusting | | | | | | Extremely disgusting |
|---|---|---|---|---|---|---|---|
| <ol> <li>Shoplifting a candy bar from a convenience store</li> </ol> | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 2. Hearing two strangers having sex | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 3. Stepping on dog poop | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 4. Stealing from a neighbor | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 5. Performing oral sex | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| <ol><li>Sitting next to someone who has red sores on their arm</li></ol> | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| <ol><li>A student cheating to get good grades</li></ol> | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| Watching a pornographic video | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| <ol><li>Shaking hands with a stranger who has sweaty palms</li></ol> | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 10. Deceiving a friend | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 11. Finding out that someone you don't like has sexual fantasies about you | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 12. Seeing some mold on old leftovers in your refrigerator | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| <ol><li>Forging someone's signature on a legal document</li></ol> | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| <ol> <li>Bringing someone you just met back to your room to have sex</li> </ol> | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| <ol><li>Standing close to a person who has body odor</li></ol> | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| <ol><li>Cutting to the front of a line to purchase the last few tickets to a show</li></ol> | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 17. A stranger of the opposite sex intentionally rubbing your thigh in an elevator | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 18. Seeing a cockroach run across the floor | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 19. Intentionally lying during a business transaction | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 20. Having anal sex with someone of the opposite sex | 0 | 1 | 2 | 3 | 4 | 5 | 6 |
| 21. Accidentally touching a person's bloody cut | 0 | 1 | 2 | 3 | 4 | 5 | 6 |

### Revised SocioSexual Orientation Inventory (Penke & Asendorpf, 2008)

Penke, L., & Asendorpf, J. B. (2008). Beyond global sociosexual orientations: A more differentiated look at sociosexuality and its effects on courtship and romantic relationships. *Journal of Personality and Social Psychology, 95*, 1113-1135.

#### Appendix

The Revised Sociosexual Orientation Inventory (SOI-R)

Please respond honestly to the following questions:

□ 5 – about once every two weeks
□ 6 – about once a week
□ 7 – several times per week
□ 8 – nearly every day
□ 9 – at least once a day

| Please respond | nonestry to | the following questio | ns: | | | | | |
|---|---|---|---|---|---|---|---|---|
| 1. With how | many differer | nt partners have you h | ad sex within | the past 12 month | hs? | | | |
| 0 | 1 | 2 | 3 | 4 | 5–6 | 7_9 | 10-19 | 20 or more |
| | many differer | nt partners have you h | _ | | | | | 20 01 111010 |
| 0 | 1 | 2 | 3 | 4 | 5-6 | 7–9 | 10-19 | 20 or more |
| 3. With how i | many differer | nt partners have you h | ad sexual inte | ercourse without h | aving an interest | in a long-term | committed relations | ship with this |
| person? | • | | | | · | | | |
| 0 | 1 | 2 | 3 | 4 | 5-6 | 7–9 | 10-19 | 20 or more |
| 4. Sex withou | t love is OK. | | | | | | | |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 |
| Strongly dis | agree | | | | | | | Strongly agree |
| <ol><li>I can imagi</li></ol> | ine myself be | ing comfortable and | enjoying "cast | al" sex with diffe | rent partners. | | | |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 |
| Strongly disag | ree | | | | | | | Strongly agree |
| 6. I do not wa | ant to have se | x with a person until | I am sure tha | t we will have a l | ong-term, seriou | s relationship. | | |
| 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 |
| Strongly disag | ree | | | | | | | Strongly agree |
| | do you have | fantasies about havin | g sex with so | meone with whom | you do not hav | e a committed re | mantic relationship | p? |
| □ 1 – never | | | | | | | | |
| □ 2 – very sel | dom | | | | | | | |
| □ 3 – about or | nce every two | or three months | | | | | | |
| □ 4 – about or | | | | | | | | |
| □ 5 – about or | | weeks | | | | | | |
| □ 6 – about or | | | | | | | | |
| □ 7 – several | | ek | | | | | | |
| □ 8 – nearly e | | | | | | | | |
| □ 9 – at least | | | | | | | | |
| | | ience sexual arousal v | when you are | in contact with so | meone with who | m you do <i>not</i> h | ave a committed ro | mantic |
| relationship | ? | | | | | | | |
| □ 1 – never | | | | | | | | |
| □ 2 – very sel | | | | | | | | |
| | | or three months | | | | | | |
| □ 4 – about or | | | | | | | | |
| □ 5 – about or | | weeks | | | | | | |
| □ 6 – about or | | | | | | | | |
| □ 7 – several | | 2K | | | | | | |
| □ 8 – nearly e | | | | | | | | |
| □ 9 – at least | | ton do vou bavo sece | tanaous factor | ios about basine | or with compan | a wan bawa inst | mat? | |
| 9. In everyday □ 1 – never | me, now on | ten do you have spon | taneous rantas | nes about naving s | sea with someon | e you have just | met: | |
| | dom | | | | | | | |
| □ 2 – very sel | | or three months | | | | | | |
| | | or three months | | | | | | |
| □ 4 – about or | nce a month | | | | | | | |

Items 1-3 should be coded as  $0=1, 1=2, \ldots, 10-19=8, 20$  or more =9; they can then be aggregated to form the Behavior facet. After Item 6 is reverse coded, Items 4-6 can be aggregated to form the Attitude facet. Aggregating Items 7-9 results in the Desire facet. Finally, all nine items can be aggregated as the total score of global sociosexual orientation.

When Items 1-3 are presented with open response format instead of the rating scales, Items 2, 4, and 7 of the original SOI (Table 1) can be added to the SOI-R to allow for calculating the SOI total score in addition to the SOI-R scores. In this case, the open responses should be recoded to the rating scale format (i.e.,  $0 = 1, 1 = 2, \ldots, 20$  to max = 9) before the SOI-R scores are determined.

Alternatively, we also developed a version of the SOI-R with 5-point rating scales, which might be more appropriate for samples with less educated or less test-experienced participants. In this version, the scale alternatives are 0, 1, 2-3, 4-7, and 8 or more for the Behavior items, 1 (strongly disagree) to 5 (strongly agree) for the Attitude items, and never, very seldom, about once a month, about once a week, and nearly every day for the Desire items. In a large, heterogeneous online sample (N = 8,549), the SOI-R with five response alternatives per item achieved good internal consistencies ( $\alpha = .83$ , .81, .82, and .85 for the total score and the facets Behavior, Attitude, and Desire, respectively). Further information on the SOI-R can be found at www.larspenke.eu/soi-r

#### Mental Health Measures

Patient Health Questionnaire (PHQ-9; Kroenke & Spitzer, 2002)

Kroenke K., Spitzer R.L. (2002). The PHQ-9: a new depression and diagnostic severity measure. *Psychiatr Ann*, 32: 509-21.

(Note: The question about suicide has been deleted).

Over the last 2 weeks, how often have you been bothered by any of the following problems? (0 = not at all; several days = 1; More than half the days = 2; Nearly every day = 3)

- 1. Little interest or pleasure in doing things
- 2. Feeling down, depressed, or hopeless
- 3. Trouble falling or staying asleep, or sleeping too much
- 4. Feeling tired or having little energy
- 5. Poor appetite or overeating
- 6. Feeling bad about yourself/failure
- 7. Trouble concentrating on things
- 8. Moving or speaking so slowly that other people could have noticed. Or being fidgety/restless.

If you checked off any problems, how difficult have these problems made it for you to do your work, take care of things at home, or get along with other people?

## PAI-BOR (Morey, 1991)

Morey, L. C. (1991). *Personality Assessment Inventory: Professional Manual.* Odessa, FL: Psychological Assessment Resources.

Read each statement and decide if it is an accurate statement about you. Circle your answer after each statement.

False, not at all true – F Slightly True – ST Mainly True – MT Very True - VT

| 1. My mood can shift quite suddenly. | F | ST | MT | VT | |
|---|---|---|---|---|---|
| 2. My attitude about myself changes a lot. | F | ST | MT | VT | |
| 3. My relationships have been stormy. | F | ST | MT | VT | |
| 4. My moods get quite intense. | F | ST | MT | VT | |
| 5. Sometimes I feel terribly empty inside. | F | ST | MT | VT | |
| 6. I want to let certain people know how much they've hurt me. | . F | ST | MT | VT | |
| 7. My mood is very steady. | F | ST | MT | VT | |
| 8. I worry a lot about other people leaving me. | F | ST | MT | VT | |
| 9. People once close to me have let me down. | F | ST | MT | VT | |
| 10. I have little control over my anger. | F | ST | MT | VT | |
| 11. I often wonder what I should do with my life. | F | ST | MT | VT | |
| 12. I rarely feel very lonely. | F | ST | MT | VT | |
| 13. I sometimes do things so impulsively that I get into trouble. | F | ST | MT | VT | |
| 14. I've always been a pretty happy person. | F | ST | MT | VT | |
| 15. I can't handle separation from those close to me very well. | F | ST | MT | VT | |
| 16. I've made some real mistakes in the people I've picked as fri | ends. F | ST | MT | VT | |
| 17. When I'm upset, I typically do something to hurt myself. | F | ST | MT | VT | |
| 18. I've had times when I was so mad I couldn't do enough to ex | kpress n | ny anger. | F | ST | MT VT |
| 19. I don't get bored very easily. | F | ST | MT | VT | |
| 20. Once someone is my friend, we stay friends. | F | ST | MT | VT | |
| 21. I'm too impulsive for my own good. | F | ST | MT | VT | |
| 22. I spend money too easily. | F | ST | MT | VT | |
| 23. I'm a reckless person. | F | ST | MT | VT | |
| 24. I'm careful about how I spend my money. | F | ST | MT | VT | |

#### Family Questionnaire (Felitti, 1997)

Felitti, V. J., Anda, R. F., Nordenberg, D., Williamson, D. F., Spitz, A. M., Edwards, V., ... & Marks, J. S. (1997). Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults: The Adverse Childhood Experiences (ACE) Study. *American journal of preventive medicine*, *56*(6), 774-786.

Please answer these questions recognitioning back to your childhood using the scale:

1 2 3 4 5
Not at All Very Often

- 1. How often did a parent or other adult in the household make you feel that you were loved, supported and cared for?
- 2. How often did a parent or other adult in the household swear at you, insult you, put you down, or act
- 3. How often did a parent or other adult in the household express physical affection for you, such as
- 4. How often did a parent or other adult in the household push, grab, shove, or slap you?
- 5. How often would you say that a parent or other adult in the household behaved violently toward a
- 6. How often would you say there as quarreling, arguing, or shouting between your parents?
- 7. How often would you say there was quarreling, arguing, or shouting between you're a parent and you?
- 8. How often would you say there was quarreling, arguing, or shouting between a parent and one of
- 9. How often would you say there was quarreling, arguing, or shouting between your sibling(s) and you?
- 10. Would you say the household you grew up in was chaotic and disorganized?
- 11. In your childhood, did you live with anyone who was a problem drinker or alcoholic, or who used street drugs?
- 12. Would you say that the household you grew up in was well-organized and well-managed?
- 13. Would you say you were neglected while you were growing up, that is, left on your own to fend for yourself?

Perceived Stress Scale (Cohen, Kamarck, & Mermelstein, 1983)

Cohen, S., Kamarck, T., & Mermelstein, R. (1983). A global measure of perceived stress. *Journal of health and social behavior*, 385-396.

0 = Never 1= Almost Never 2=Sometimes 3=Fairly Often 4=Very Often

#### In the last month:

- 1. How often have you been upset because of something that happened unexpectedly?
- 2. How often have you felt that you were unable to control the important things in your life?
- 3. How often have you felt nervous and "stressed"?
- 4. How often have you felt confident about your ability to handle your personal problems?
- 5. How often have you felt that things were going your way?
- 6. How often have you found that you could not cope with all the things you had to do?
- 7. How often have you been able to control irritations in your life?
- 8. How often have you felt that you were on top of things?
- 9. How often have you been angered because of things that were outside of your control?
- 10. How often have you felt difficulties were piling up so high that you could not overcome them?